CLINICAL TRIAL: NCT00925093
Title: Antibiotics in Cerebrospinal Fluid Following Intravenous Injection
Brief Title: Study of Antibiotics in Cerebrospinal Fluid Following Intravenous Injection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary investigator left institution
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Morten Gustav Poulsen, MD, Aarhus University Hospital, Aarhus Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AUH-MGP-AB-CSV-2009-1
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2009-06

CONDITIONS: Neurosurgery
Keywords: vancomycin; teicoplanin; linezolid; intravenous; cerebrospinal fluid; CSF; pharmacokinetics; penetration; blood-brain barrier; Pharmacokinetics of three antibiotics in relation to cerebrospinal fluid
MeSH Terms: interventions — Vancomycin; Teicoplanin; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vancomycin (Active Comparator): Vancomycin is administered intravenously and subsequently measured in cerebrospinal fluid sample
  Interventions: Drug: Vancomycin
- Teicoplanin (Active Comparator): Teicoplanin is administered intravenously and subsequently measured in cerebrospinal fluid sample
  Interventions: Drug: Teicoplanin
- Linezolid (Active Comparator): Linezolid is administered intravenously and subsequently measured in cerebrospinal fluid sample
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Vancomycin — Vancomycin is administered intravenously and subsequently measured in cerebrospinal fluid sample
  Arms: Vancomycin
Drug: Teicoplanin — Teicoplanin is administered intravenously and subsequently measured in cerebrospinal fluid sample
  Arms: Teicoplanin
Drug: Linezolid — Linezolid is administered intravenously and subsequently measured in cerebrospinal fluid sample
  Arms: Linezolid

SUMMARY:
Three different antibiotics are used to prevent infection in case of neurosurgery - this study examines to which extent the antibiotics penetrate from the blood to the cerebrospinal fluid (surrounding the brain).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Already having an external CSF drain
* Scheduled for neurosurgery requiring antibiotic prophylaxis (most commonly placement of an internal drain ("shunt")

Exclusion Criteria:

* Infection or colonization requiring other than standard prophylactic antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of antibiotics in cerebrospinal fluid | 1, 2, 4, 6, 12 hours
  Concentration in CSF past i.v. injection